CLINICAL TRIAL: NCT06222801
Title: Open Prospective Observational Cohort Study of the Effectiveness and Safety of Cytokinogenetic Therapy in Patients With Cancer Based on TCTD-1 Patient Registry
Brief Title: The 1st Tumor CytokinoTherapy Database (TCTD-1)
Status: Recruiting | Type: Observational
Sponsor: OncoCareClinic 308 Ltd (Other)
Responsible Party: Sponsor
Other Study IDs: REF.AND.ING 2022
Record Dates: First submitted 2023-12-29; First posted 2024-01-25 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-01

CONDITIONS: Oncology
Keywords: TNF-α; Tumor necrosis factor alpha; interferon gamma; IFN-γ; Cancer; Cytokinogenetic therapy
MeSH Terms: conditions — Neoplasms | interventions — Tumor Necrosis Factor-alpha; Interferon-gamma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tumor necrosis factor alpha — Antitumor agent. Immunomodulatory agent.
  Other Names: TNF-α; Refnot
Drug: Interferon gamma — Immunostimulating agent.
  Other Names: IFN-γ; Ingaron

SUMMARY:
Predicting the response of patients diagnosed with cancer to cytokinotherapy is essential to guide anti-tumor therapy complex strategy and subsequent adjuvant approach. Cytokinotherapy is a cost-effective, well-known available method of therapy for the patients with tumors. The objective response possibly correlates to the tumor's size, aggressiveness, age, and other primary factors. Multifactor analysis requires a large amount of data. Therefore, the investigators created the first database aimed to collect data concerning the patients with cancer and the clinical outcomes of cytokinogenetic therapy. The acquired data must be processed to detect the key factors effecting the outcomes. Cytokinotherapy is a universal therapeutic approach, although we lack information that would help to personalize it and reduce the rate of progression. The main goal is to find the relationship between initial patients' characteristics and effectiveness of cytokinotherapy for early risks detection. The predictive models that could be elaborated from the TCTD-1 analysis will complement knowledge of cytokinotherapy rationale. Predicting survival or other significant clinical criteria using TCTD-1 analysis results would greatly benefit the cancer patients' management.

DETAILED DESCRIPTION:
The investigators plan to carry out an open prospective observational cohort study during 10 years based on TCTD-1 registry of patients with cancer diagnoses in order to assess the effectiveness and safety of cytogenetic therapy. Demographic, clinical, radiological, genetical and laboratory variables (TNF alpha) will also be collected. OS will be defined as the time elapsed between the application for cytogenetic therapy with cancer diagnosis and the patient's death.

Objectives:

1. To establish a longitudinal observational registry of patients with cancer based on clinical and laboratory analytical variables.
2. To identify the patients with a high potential of cytokinogenetic therapy and/or low risk of complications.
3. To assess the effectiveness and safety of cytogenetic therapy in patients with cancer.
4. To determine the relationship between the initial patients' features and effectiveness and safety criteria (objective response, overall survival, AE rate, etc.).
5. To develop a predictive model.
6. To validate the model and compare it with currently available predictive models.

   The methodological properties of the study are described below:
7. - Type of design Open prospective observational registry study.
8. - Study population Patients diagnosed with neoplasia with an indication for cytogenetic therapy.
9. - Inclusion and exclusion criteria Adult patients aged 18 years or older with cancer who do not meet exclusion criteria, applied to the OncoCare308 Clinic Ltd. hospital for cytogenetic therapy, and are eligible to complete or have completed at least one course of cytogenetic therapy, as determined by the site, who do not meet any exclusion criteria.
10. -The study exclusion criteria are:

    * Patients under 18 or over 95 years
    * Patients with hematologic cancer or thyroid tumors
    * Patients with contraindications for cytogenetic therapy
    * Patients who die before the start of therapy or before the first course completeness
    * Patients who do not sign the informed consent to be enrolled under the clinical observation in the hospital
11. - Sample size The purpose of the study is to recruit as many patients as possible among those who wish to participate.
12. - Recruitment Once the enrollment criteria have been assessed, each patient will be assigned a unique code that will be used to anonymously manage any of the information obtained during the study. Thus, the confidentiality of the data will be guaranteed at all times from the moment of recruitment.
13. - Intervention Not applicable.
14. - Follow up The patient will be monitored for at least 4 years up to 10 years, compiling all the specific variables of this study and the possible complications and mortality that occurred in this period.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged 18 years or older with cancer who do not meet exclusion criteria, applied to the OncoCare308 Clinic Ltd. hospital for cytogenetic therapy, and are eligible to complete or have completed at least one course of cytogenetic therapy, as determined by the site.

Exclusion Criteria:

* Patients under 18 or over 95 years
* Patients with hematologic cancer or thyroid tumors
* Patients with contraindications for cytogenetic therapy
* Patients who die before the start of therapy or before the first course completeness
* Patients who do not sign the informed consent to be enrolled under the clinical observation in the hospital

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an oncological diagnosis and an indication for cytokinogenetic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2032-09-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 10 years
  Number of objective responses to therapy before progression or relapse.

SECONDARY OUTCOMES:
Changes in functional status since the start of cytokinegenetic therapy during treatment and observation. | 10 years
  The Karnofsky index parameter will be evaluated.
Overall survival of patients since the start of cytokinogenetic therapy. | 10 years
  The time elapsed between the start of cytogenetic therapy and the death of the patient (for any reason, including those not related to oncology).
Relapse-free survival of patients since the start of cytokinogenetic therapy. | 10 years
  The time elapsed between the start of cytokinogenetic therapy and the detection of relapse or death of the patient (for any reason, including those not related to oncology).
The appearance of toxicity from the moment of initiation of cytokinogenetic therapy. | 10 years
  AEs associated with cytokine therapy.
Changes in the level of TNF in the blood since the start of cytokinegenetic therapy during treatment and observation. | 10 years
  Dynamics of TNF levels in the blood throughout the study.
Duration of response to cytokinogenetic therapy. | 10 years
  Duration of response to therapy as time to event (progression or relapse). Analysis of duration of response will be performed in the group of patients who responded to therapy.
Disease control rate. | 10 years
  The number of patients who achieve disease control will be assessed every 3 months until progression or relapse occurs.

CONTACTS AND LOCATIONS:
Locations (1):
- OncocareClinic 308, Moscow, Russia